CLINICAL TRIAL: NCT02752295
Title: Intensive Stress Coping Intervention Week - A Secondary Prevention For Real World Affective Disorder Patients
Acronym: ISCIW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Sanatorium Hera Vienna (Unknown)
Responsible Party: Principal Investigator, Robert Winker, Prim.Priv. Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ISCIW trial
Record Dates: First submitted 2016-04-07; First posted 2016-04-26 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Affective Disorders; Psychological Stress; Inflammation; Oxidative Stress; Anxiety Disorders; Mood Disorders; Emotions
MeSH Terms: conditions — Mood Disorders; Stress, Psychological; Inflammation; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Waiting list, intervention after EOS (No Intervention): control group / waiting list one week stress-coping intervention planned after end of study (EOS) without one week stress-coping intervention AND without an additional two days follow-up care
- Stress-coping week without follow-up (Active Comparator): active comparator with one week stress-coping intervention BUT without an additional two days follow-up weekend
  Interventions: Behavioral: stress-coping week
- Stress-coping week with follow-up (Active Comparator): active comparator with one week stress-coping intervention AND with an additional two days follow-up weekend
  Interventions: Behavioral: stress-coping week; Behavioral: additional two days follow-up weekend

INTERVENTIONS:
Behavioral: stress-coping week — The multidisciplinary team will offer Mindfulness-Based Stress Reduction (MBSR), group psychotherapy (resilience, Cognitive Behavioral Analysis System of Psychotherapy CBASP, psychodynamic therapy), relaxation training, nutrition course, stress-coping and physical training in a group setting.
  Arms: Stress-coping week with follow-up; Stress-coping week without follow-up
Behavioral: additional two days follow-up weekend — A two-days follow-up which recapitulates previous treatment elements.
  Arms: Stress-coping week with follow-up

SUMMARY:
This study intents to determine who will benefit from an intensive brief stress coping intervention week (ISCIW) as secondary prevention for real world affective disorder patients.

DETAILED DESCRIPTION:
Affective disorders are associated with a substantial personal and socio-economic burden. This study evaluates an intensive brief stress-coping intervention week (ISCIW) as feasible follow-up treatment for real world patients who suffer from this highly prevalent and chronic stress-related disorders. Stress-associated blood (Interleukin-6, Homocystein, Myeloperoxidase), saliva cortisol and psychosocial screening parameters will be analyzed to determine who will benefit from the ISCIW. All patients were identified in a preventive medical screening before pre-treatment for at least three month as outpatient and the following inclusion to the follow-up ISCIW-trial at the Health and Prevention Center, Sanatorium Hera, Vienna, Austria. For the three planed groups and interventions see interventions and arms.

ELIGIBILITY:
Inclusion Criteria:

* Affective or anxiety disorder DSM-IV diagnosis (structured interview, M.I.N.I. International Neuropsychiatric Interview )
* Minimum 3-weeks previous therapeutic treatment as outpatient at the Health and Prevention Center, Sanatorium Hera, Vienna, Austria
* Clinical Global Impression - Severity (CGI-S) score > 2 points
* Minimum improvement of 1 CGI-S points as outpatient
* Written informed consent

Exclusion Criteria:

* More than 60 days away sick per year in the last year before intervention
* Therapy adherence as outpatient at the Health and Prevention Center, Sanatorium Hera, Vienna, Austria
* Work Ability Index (WAI) score < 25 points
* Major neurological or cognitive deficits
* Current psychotic symptoms
* Current or previous DSM-IV diagnosis of substance dependence, except for nicotine or current substance abuse
* Failures to comply with the study protocol or to follow the instructions of the study team
* Currently requested application for retirement
* Middle to high suicidal tendency in the M.I.N.I.-examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change of saliva cortisol | Change from baseline saliva sample at week 1 to end of study visit at week 38

SECONDARY OUTCOMES:
Change of myeloperoxidase | Change from baseline at week 1 to end of study visit at week 38
Change of interleukin-6 | Change from baseline at week 1 to end of study visit at week 38
Change of homocystein | Change from baseline at week 1 to end of study visit at week 38
Change of psychometric stress-index (Questionnaire) | Change from baseline at week 1 to end of study visit at week 38

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pilger A, Haslacher H, Ponocny-Seliger E, Perkmann T, Bohm K, Budinsky A, Girard A, Klien K, Jordakieva G, Pezawas L, Wagner O, Godnic-Cvar J, Winker R. Affective and inflammatory responses among orchestra musicians in performance situation. Brain Behav Immun. 2014 Mar;37:23-9. doi: 10.1016/j.bbi.2013.10.018. Epub 2013 Oct 26. PMID 24513877